CLINICAL TRIAL: NCT05116917
Title: Nivolumab, Ipilimumab and Radiation in Combination With Influenza Vaccine in Patients With Pancreatic Cancer (INFLUENCE)
Brief Title: Immunotherapy Combined With Radiation and Influenza Vaccine for Pancreatic Cancer.
Acronym: INFLUENCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the precpecified interim analysis the predictive probability was below 10% for the prespecified endpoint.
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Inna Chen, MD, Principal Investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 2118
Record Dates: First submitted 2021-10-23; First posted 2021-11-11 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Check point inhibitors; Influenza vaccine
MeSH Terms: conditions — Pancreatic Neoplasms; Influenza, Human | interventions — Nivolumab; Ipilimumab; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in the study to treatment with nivolumab, ipilimumab and radiation in combination with influenza vaccine, until 30 participants have been treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): SBRT of 15 Gy will be given on day 1 of the first cycle. Nivolumab 3 mg/kg (up to 240 mg maximum) will be given on day 1 (± 3 days) of each 14-day treatment cycle until the progression of disease or maximum of 48 weeks, discontinuation due to toxicity, withdrawal of consent. Ipilimumab 1 mg/kg will be given on day 1 cycle 1 (± 3 days) and once more after 6 weeks. Nivolumab will be administered as an IV infusion over 60 (± 5) minutes and then, after a 30 minutes rest period, ipilimumab will be administered as an IV infusion over 30 (± 5) minutes. Seasonal influenza vaccine is given IM or via PharmaJet Stratis Needle-Free Injection System, 0.5 mL per dose as a single on day 1 cycle 1 (± 3 days).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Biological: Influenza vaccine; Radiation: SBRT

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg (up to 240 mg maximum) will be given on day 1 (± 3 days) of each 14-day treatment cycle
  Other Names: Opdivo®
Drug: Ipilimumab — 1 mg/kg will be given on day 1 cycle 1 (± 3 days) and once more after 6 weeks
  Other Names: Yervoy®
Biological: Influenza vaccine — Seasonal influenza vaccine is given IM or via PharmaJet Stratis Needle-Free Injection System, 0.5 mL per dose as a single on day 1 cycle 1 (± 3 days)
Radiation: SBRT — * A total dose of 15 Gy as a single fraction is prescribed as the mean dose to the PTV.
  * PTV should be covered by 95% isodose (PTV D99% > 95%).

SUMMARY:
Pancreatic cancer (PC) remains a dreadful disease due to its often advanced stage at diagnosis and poor sensitivity to chemotherapy. Progression after 1. line chemotherapy is inevitable in patients with advanced PC, and treatment options for patients who progress after 1. line chemotherapy are limited. Considering the emerging role of the tumor microenvironment, the combination of checkpoint blocking antibodies with immunomodulation of the tumor microenvironment could lead to better responses in tumor historically resistant to radiation and checkpoint blocking antibody approaches as single modalities. Influenza vaccination in cancer patients receiving immune checkpoint inhibitors resulted in a better survival, irrespective of the anticancer treatment outcome. Influenza vaccine facilitates both T- and B cell activation and drives interferon-gamma response, supporting the rationale for combining of influenza vaccine with immune checkpoint inhibition and radiation (NCT02866383).

Based on these considerations, the proposed treatment with SBRT of 15 Gy in combination with nivolumab, ipilimumab and influenza vaccine may have the potential to provide meaningful clinical benefit by generating durable clinical responses, thereby improving quality of life (QoL) and potentially extending survival.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is the fourth leading cause of cancer death, and each year 1000 Danes are diagnosed with PC, 80% of which are advanced stage. Survival rates are meager, currently approaching 10% at 5 years postdiagnosis, and have scarcely improved over the last 50 years. PC is highly resistant to conventional treatments, and nearly all patients develop metastases and die. As the incidence of PC continuously rises while treatment response rates remain incredibly low, a lack of effective therapy options and accurate predictive biomarkers is a real cause for concern and underlines the need for further research in this area.

Immunotherapy has not been successful in PC patients primarily due to a lack of pre-existing T-cell immunity and/or a highly immunosuppressive tumor microenvironment. "Non-immunogenicity" of PC with high prevalence of immunosuppressive cells and typically a scarcity of tumor-infiltrating effector lymphocytes is considered as one of the reasons for lacking responsiveness to single-agent immunotherapies. Considering the emerging role of the tumor microenvironment, the combination of checkpoint blocking antibodies with immunomodulation of the tumor microenvironment could lead to better responses in tumor historically resistant to radiation and checkpoint blocking antibody approaches as single modalities. Preliminary data from the phase 2 study CHECKPAC (NCT02866383) showed durable clinical benefit in a small subgroup of patients after the addition of stereotactic body radiation therapy (SBRT) of 15 Gy to the combination of nivolumab and ipilimumab (Herlev internal data) in patients with resistant metastatic PC.

Influenza vaccination in cancer patients receiving immune checkpoint inhibitors inexplicably was associated with a better survival, irrespective of the anticancer treatment outcome. Influenza vaccine facilitates both T- and B cell activation and drives interferon-gamma response, supporting the rationale for combining of influenza vaccine with CHECKPAC strategy. Based on these considerations, the proposed treatment with nivolumab, ipilimumab and radiation in combination with influenza vaccine may potentially provide meaningful clinical benefit by generating durable clinical responses, thereby improving quality of life (QoL) and potentially extending survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histological or cytological confirmation of advanced pancreatic carcinoma prior to entering this study
* Prior therapy requirements:

  * There is no upper limit on the number of prior chemotherapy regimens received. Participants must have received and progressed during or after at least 1 line of systemic chemotherapy in the metastatic setting (gemcitabine or 5-FU based regimens).
  * Notes:

    * If a participant received adjuvant/neoadjuvant systemic combinational therapy, and progressed within 6 months, the adjuvant/neoadjuvant treatment will be considered as 1 line of systemic treatment.
    * In general, discontinuation of 1 drug in a multi-drug regimen and continuation of other drug(s), is considered part of the same line of treatment. Restarting the same regimen after a drug holiday or maintenance chemotherapy can also be considered part of the same line of treatment. Switching from IV (5-FU) to an oral formulation (capecitabine) of the same drug is also considered part of the same line of treatment
    * Minimum time from first systemic therapy for recurrent/metastatic adenocarcinoma of pancreas to progression should be at least 3 months
* Age 18 years and older
* ECOG/WHO Performance Status (PS) 0-1
* All participants will be required to undergo mandatory pre- and on-treatment biopsies at acceptable clinical risk as judged by the investigator. An archival pre-treatment sample is not acceptable.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
  * Platelet count ≥ 75 x 10⁹/L
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * AST/ALT ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP) must use method(s) of contraception as indicated in Appendix 3. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. WOCBP should therefore use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab is up to 25 days. Men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Subjects must have signed and dated a BIOPAC approved written informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Current or prior use of immunosuppressive medication within 14 days before the first dose of nivolumab, ipilimumab and radiation in combination with influenza vaccine. The following are exceptions to this criterion:

  * Intranasal, inhaled, or topical steroids; or local steroid injections (e.g. intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Participants should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* Already received the influenza vaccine for the current season of inclusion
* WOCBP who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
  ORR in all patients using Investigator assessments

SECONDARY OUTCOMES:
Duration of response (DoR) | 12 months
  DoR in all patients using Investigator assessments according to RECIST 1.1.
Disease control rate (DCR) | 12 months
  DCR in all patients using Investigator assessments according to RECIST 1.1.
Progression free survival (PFS) | 12 months
  PFS in all patients using Investigator assessments according to RECIST 1.1.
Overall survival (OS) | 12 months
  OS in all patients using Investigator assessments according to RECIST 1.1.
EORTC QLQ-C30 | 12 months
  Adjusted mean change from baseline in global QoL
Treatment-related adverse events as assessed by CTCAE v5.0 | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Inna M Chen, Principal Investigator — Herlev Sygehus
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No